CLINICAL TRIAL: NCT06249360
Title: Influence of Lymphatic System Reflux After Operation in Patients With Lymphatic Disease
Brief Title: Lymphatic System Reflux After Lymphatic Operation
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301216B0
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-08

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Limb Lymphedema: Patients with cancer-related unilateral lower limb lymphedema were enrolled.
  Interventions: Other: Veins with reflux; Other: Reflux-free recipient veins

INTERVENTIONS:
Other: Veins with reflux — This group included patients who used only recipient veins with reflux
Other: Reflux-free recipient veins — This group included patients who utilized only reflux-free recipient veins

SUMMARY:
This study aimed to determine the impact on outcomes when recipient veins with reflux were used for LVA for the treatment of unilateral lower limb lymphedema.

DETAILED DESCRIPTION:
The use of recipient veins with reflux for lymphaticovenous anastomosis (LVA) is discouraged because of the common belief that it may lead to venous-lymphatic reflux (VLR), a phenomenon in which venous blood is refluxed into the lymphatic lumen after anastomosis, which can lower the long-term patency rate. However, this concept has yet to be validated.

ELIGIBILITY:
Inclusion Criteria:

* This study including patients diagnosed with lymphatic-related diseases at Kaohsiung Chang Gung Memorial Hospital from October 1, 2015, to December 31, 2022.
* Patients who underwent LVA for unilateral lower-limb lymphedema.

Exclusion Criteria:

* Patients under the age of 20.
* Patients lost to follow-up or with incomplete data.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (age >20 years) receiving LVA for lower limb lymphedema at a tertiary medical center were retrospectively reviewed from October 2015 to December 2022.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Volume change after LVA. | 6/12 months
  The primary endpoint was the volume change at 6/12 months after LVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan